CLINICAL TRIAL: NCT06696053
Title: Hospital and Extra-hospital Nursing Care for Tuberculosis
Acronym: FOLLOWTUB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP240272; IDRCB-2024-A01634-43 (Other: ANSM)
Record Dates: First submitted 2024-11-18; First posted 2024-11-19 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; education nursing program
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Tuberculosis (Experimental)
  Interventions: Other: Transversal therapeutic education

INTERVENTIONS:
Other: Transversal therapeutic education — Additional patient consultation for therapeutic education with nurses.

SUMMARY:
The incidence of tuberculosis has decreased over the last 2 years on the national territory (6.4/100,000 inhabitants) but remains twice as high in Ile de France where it is increasing with an increase of almost 10% in the number of cases. reported between 2015 and 2017 . the notification rate of tuberculosis disease for the year 2020 was 14.3 cases per 100,000 inhabitants (i.e. 1757 cases declared) which is more than double that found at the national level . As the disease is multifocal, patients are likely to be hospitalized in different departments with variable care and compliance support offered. One of the major issues is compliance with treatment. Indeed, INVS data (2008-2014) report a percentage of treatment completed in pulmonary tuberculosis of 73% . Among these cases, 20% had a potentially unfavorable outcome, including 45% lost to follow-up, which creates a risk of relapse and contagiousness for those around them. The latest data reported in 2022 over the period 2014-2018 seem to show an increase in treatment completeness but completeness remains variable from one region to another and from one year to another Using Public Health France data, the investigator were able to collect the proportion of completeness of treatment at Saint Antoine hospital, which is 60% over the period 2014-2016 (Public Health France, unpublished data). In more recent work carried out within the department retrospectively between 2019-2021, the investigator compared treatment outcomes depending on whether or not patients benefit from ETP support and it is 66% among patients without it. benefited, thus confirming the data from Public Health France over a more recent period.. In this context, several other studies have shown the interest of a therapeutic education program on the completeness of the treatment.

DETAILED DESCRIPTION:
As part of a pilot study, our objective is to evaluate the benefit of a transversal therapeutic education nursing program within an AP-HP hospital in order to significantly increase the number of patients who have followed their entire treatment as recommended by the WHO Our main objective is to Evaluate the impact of a transversal therapeutic education nursing program on the outcome rate of completed anti-tuberculosis treatment in patients diagnosed with tuberculosis disease at St Antoine hospital.

The design of the study is Prospective, multicenter pilot study evaluating the impact of a transversal therapeutic education nursing program on the completeness of treatment with comparison on historical data.

40 patients over 12 months for all centers will be enroled No interim analysis was planned The analysis will be carried out at the end of the research after freezing the database, with the SAS V9.4 software.

Patient characteristics will be described by the number and proportion for qualitative variables and by their median and interquartile range for continuous variables.

The outcome rate of completed anti-tuberculosis treatment will be calculated as well as its 95% confidence interval (exact Clopper-Pearson method) and compared to the theoretical proportion of 60% by an asymptotic Wald test. A patient lost to follow-up will be considered a failure.

ELIGIBILITY:
Inclusion Criteria:

* Patient for whom a diagnosis of tuberculosis disease or latent tuberculosis according to the recommendations of the IDSA / CDC has been made and treatment with antituberculosis drugs started less than 3 weeks ago (9)
* Patient followed in one of the participating departments of the St Antoine hospital (internal medicine, rheumatology, gastroenterology, hepatology, geriatrics)
* Patient having signed informed consent
* Patient whose age > 18 years
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of outcomes of completed antituberculosis treatment | At 6, 9 and 12 month post inclusion
  A favorable treatment outcome will be defined by a composite criterion, namely: treatment compliance > 80% (self-questionnaire during visits), 80% of visits honored and clinical cure for the referring physician.

SECONDARY OUTCOMES:
Rate of patients lost to follow-up among patients included | At 6 and 12 month post inclusion
Rate of caregivers showing an improvement in their knowledge before and after the implementation of the training and information action on tuberculosis | At inclusion and at 12 month
  via questionnaires
Rate of patients showing improvement in their knowledge before and after the implementation of the training and information action on tuberculosis | At inclusion visite,1, 6, 9 and 12 months after inclusion
  via questionnaires
Evolution of patients' quality of life before and at the end of treatment | At inclusion visite,1, 6, 9 and 12 months after inclusion
  SF36 scale
Caregivers' program satisfaction scale | At inclusion visit and at 12 month
  via questionnaires
Patient Program Satisfaction Scale | At inclusion visite,1, 6, 9 and 12 months after inclusion
Number of meetings of the network for monitoring the most vulnerable patients between the city and the hospital involving the Samu social coordinated by the infectious diseases department | through the study completion and up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Emma TORRES, Nurse, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service des Maladies Infectieuses et Tropicales, Hôpital Saint-Antoine, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No